CLINICAL TRIAL: NCT04046887
Title: Phase I Study of Lonsurf in Combination With Gemcitabine and Nab-Paclitaxel in Patients With Advanced Pancreatic Ductal Adenocarcinoma (PDAC)
Brief Title: Study of Lonsurf in Combination With Gemcitabine and Nab-Paclitaxel in Patients With Advanced (PDAC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to proceed due to Neulasta difficulties and other complications.
Sponsor: Patrick Joseph Loehrer Sr. (Other)
Collaborators: Indiana University (Other); Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Patrick Joseph Loehrer Sr., Distinguished Professor of Medicine, Indiana University
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IUSCC-0664
Record Dates: First submitted 2019-08-01; First posted 2019-08-06 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Pancreatic Cancer; Pancreatic Ductal Adenocarcinoma
Keywords: Pancreatic Ductal Adenocarcinoma; Pancreatic Cancer; Metastatic Pancreatic Cancer; Locally Advanced Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — trifluridine tipiracil drug combination; Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Intervention Model Description: Initially 3 patients will be enrolled to the starting cohort. If 1 of 3 patients experience a dose-limiting toxicity (DLT) in the first cycle, then an additional 3 evaluable patients will be accrued to that dose level. Dose reductions are not permitted during cycle 1. If 2 or more patients in a cohort experience a DLT, then the previous dose will be considered the recommended phase 2 dose (PR2D) and dose escalation will terminate. Dose escalation will proceed according to the scheme above only after all patients (3 or 6 evaluable patients, depending on the incidence of DLT) have been followed for at least 1 full cycle.
  Once dose escalation has been completed, if only 2 dose levels were used to determine the RP2D and depending on how many patients were replaced, additional patients will be enrolled at the RP2D in order to obtain data for 18 patients total.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination of lonsurf + gemcitabine + nab-paclitaxel (Experimental)
  Interventions: Drug: Lonsurf; Drug: Gemcitabine; Drug: Nab-Paclitaxel

INTERVENTIONS:
Drug: Lonsurf — Lonsurf will be administered orally twice a day on days 2-6 and 16-20 of every 28-day cycle at a dose of 25 mg/m2, 20 mg/m2 or 30 mg/m2 depending on cohort assignment.
Drug: Gemcitabine — Gemcitabine will be intravenously administered on Days 1 and 15 of every 28-day cycle at a dose of 800 mg/m2, 600 mg/m2 or 1000 mg/m2 depending on cohort assignment.
Drug: Nab-Paclitaxel — Nab-Paclitaxel will be intravenously administered on Days 1 and 15 of every 28-day cycle at a dose of 100 mg/m2, 75 mg/m2 or 125 mg/m2 depending on cohort assignment.

SUMMARY:
The purpose of this study is to determine the recommended phase 2 dose (RP2D) of the combination of lonsurf, gemcitabine and nab-paclitaxel in Pancreatic ductal adenocarcinoma (PDAC)

DETAILED DESCRIPTION:
This is a single-institution, prospective, phase I dose escalation trial of lonsurf combined with gemcitabine and nab-paclitaxel using the 3+3 design. This study will enroll 18 patients over 12-15 months.

Primary Objective To determine the recommended phase 2 dose (RP2D) of the combination of lonsurf, gemcitabine and nab-paclitaxel

Secondary Objectives

1. Examine safety and toxicity of the combination
2. Estimate response rate to the combination
3. Estimate median overall survival (mOS) of the treated population
4. Estimate median progression free survival (mPFS) of the treated population
5. Estimate disease control rate (DCR) at 8 weeks
6. Evaluate quality of life while receiving the combination therapy

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old at the time of informed consent
2. Ability to provide written informed consent and HIPAA authorization
3. Untreated locally advanced Pancreatic Ductal Adenocarcinoma (PDAC) as defined by National Comprehensive Cancer Network (NCCN) guidelines or, untreated metastatic PDAC (prior adjuvant therapy is permitted if it's been greater than 6 months since completion)
4. Histologically or cytologically confirmed PDAC
5. Confirmed PDAC that is measurable or evaluable per RECIST 1.1
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
7. Gastrointestinal symptoms (nausea, vomiting, and diarrhea) of Grade 1 or less
8. Adequate organ function as defined by:

   1. Aspartate transaminase (AST) and alanine transaminase (ALT) levels ≤ 2.5 x upper limits of normal (ULN)
   2. Total bilirubin level ≤ 1.5 x ULN
   3. Creatinine level < 1.0 x ULN or creatinine clearance > 60 mL/min/1.73 m2 for patients with creatinine levels above or below the institutional normal (as determined by Cockcroft-Gault equation). For patients with a Body Mass Index (BMI) > 30 kg/m2, lean body weight should be used to calculate the glomerular filtration rate (GFR).
   4. Hemoglobin (Hgb) ≥ 9 g/dl
   5. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   6. Platelets ≥ 100 x 109/L
   7. Acceptable coagulation studies as demonstrated by prothrombin time (PT) within normal limits (+/-15%) unless they are on anticoagulation therapy
9. Life expectancy estimated at ≥ 3 months
10. Women of childbearing potential definition (WOCBP) must have a negative serum or urine pregnancy test performed within 14 days prior to initiation of study treatment.

    Any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) is classified as WOCBP if she meets the following criteria:
    1. Has not undergone a hysterectomy or bilateral oophorectomy; or
    2. Has not been naturally postmenopausal for at least 24 consecutive months (i.e. has had menses at any time in the preceding 12 consecutive months).
11. WOCBP and men must agree to use adequate contraception prior, to study entry, for the duration of study participation, and 8 weeks after the end of treatment.

Exclusion Criteria:

1. Neuropathy > Grade 1 at baseline
2. Prior systemic chemotherapy for any other malignancy (aside from adjuvant therapy for PDAC) in the last 3 years
3. Active malignancy other than PDAC (other than adequately treated cervical or vulvar carcinoma in situ, treated basal cell or squamous carcinoma of the skin, superficial bladder tumors (Ta, Tis & T1), ductal carcinoma in situ (DCIS) of the breast and low grade prostate cancer. Any cancer curatively treated >3 years prior to entry with no clinical evidence of recurrence is permitted)
4. Prior exposure to nab-paclitaxel, paclitaxel, or other taxanes
5. History of bowel obstruction in the preceding 3 months of therapy, including gastric outlet obstruction related to PDAC
6. Large, uncontrolled ascites requiring paracentesis
7. Major surgery, other than diagnostic or laparoscopic surgery, within 4 weeks prior to first dose. (Port placement would not be considered a surgery.)
8. Any known untreated brain metastases including leptomeningeal metastases
9. Pregnant or breastfeeding
10. Significant gastrointestinal disorder(s) that would, in the opinion of the Principal Investigator, prevent absorption of an orally available agent (e.g., Crohn's disease, ulcerative colitis, extensive gastric resection, and small intestinal resection)
11. Uncontrolled chronic diarrhea > Grade 1 at baseline.
12. Uncontrolled intercurrent illness including, but not limited to uncontrolled active infection, clinically significant non-healing or healing wounds, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, significant pulmonary disease, uncontrolled infection, or psychiatric illness/social situations that would limit compliance with study requirements.
13. Interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
14. History of posterior reversible encephalopathy syndrome
15. Enrollment on any additional investigational agent study
16. Known hypersensitivity to gemcitabine or taxanes
17. Significant cardiac disease including the following: unstable angina, New York Heart Association class III-IV congestive heart failure, myocardial infarction < 6 months prior to study enrollment
18. History of hemolytic-uremic syndrome
19. Known infection with Human Immunodeficiency Virus (HIV) and/or active infection with hepatitis B or hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Frequency of Dose Limiting Toxicities (DLTs) | 28 days (Cycle 1)
  Number of DLTs observed

SECONDARY OUTCOMES:
Frequency of adverse events in the safety evaluable population | from start of treatment until 30 days after treatment discontinuation (i.e up to 2 years)
  safety and toxicity data will be assessed using NCI CTCAE v5.0
Response rate to the combination of lonsurf, gemcitabine, and nab-paclitaxel in the efficacy evaluable population | from start of treatment until treatment discontinuation (i.e. up to 2 years)
  Using RECIST 1.1
Median Overall Survival (mOS) of the treated population | from start of treatment until death or last known follow up (i.e up to 2 years)
Median Progression-free Survival (mPFS) of the treated population | from start of treatment until disease progression or last follow up (i.e. up to 2 years)
Disease control rate (DCR) | 8 weeks
  Disease control rate (DCR) as defined by (complete response + partial response + stable disease)
European Organization for Research and Treatment of Cancer quality of life questionnaire | Day 1 of each cycle(each cycle is 28 days),from start of treatment until disease progression or discontinuation of treatment (i.e. up to 2 years)
  Scale scores were calculated by averaging items within scales and transforming average scores linearly. All of the scales range in score from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning whereas a high score for a symptom scale or item represents a high level of symptomatology or problems.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J Loehrer, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Melvin & Bren Simon Cancer Center, Indianapolis, Indiana, United States